CLINICAL TRIAL: NCT03210467
Title: The Changes of Plasmacytoid Dendritic Cells Frequency and Function During Pegylated Interferon α-2a and Entecavir(ETV) Treatment in Patients With Chronic Hepatitis B.
Brief Title: The Changes of Plasmacytoid Dendritic Cells Frequency and Function During Antiviral Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY011
Record Dates: First submitted 2017-06-30; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis B Infection
Keywords: chronic hepatitis B; hepatitis B virus; Pegylated Interferon α-2a; entecavir; Plasmacytoid Dendritic Cells
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- experimental group: patients who were untreated ever in immune-active phase were given subcutaneous injection of Peginterferon Alfa-2a with starting dose of 180 mg/weekly till 48 weeks.
- control group: patients who were untreated ever in immune-active phase took entecavir(ETV) for maintenance treatment.

SUMMARY:
Pegylated interferon(IFN) α-2a(Peg-IFN-α) not only inhibit viral replication, but also play an important role in immune regulation, while entecavir(ETV) drugs only inhibit viral replication. In hepatitis B infection, Plasmacytoid Dendritic Cells（pDCs） are the main effector cells in early antiviral innate immune response. This study was aimed at investigating the changes of pDCs frequency and function, and the expression of costimulatory molecules CD86(Cluster of Differentiation antigen 86) during Peg-IFN-αand entecavir(ETV) therapy.Meanwhile, investigators want to verify whether Peg-IFN-α suppressed the virus and the reduction of virus led to the recovery of pDCs function, or Peg-IFN-α enhanced pDCs function which gave rise to the decline of the virus.

DETAILED DESCRIPTION:
Pegylated interferon α-2a(Peg-IFN-α)and entecavir(ETV) drugs can inhibit viral replication , but Peg-IFN-α also play an important role in immune regulation . In hepatitis B infection, Plasmacytoid Dendritic Cells (pDCs) are the main effector cells in early antiviral innate immune response.Peg-IFN-α recommended as the first-line treatment has a higher chance to achieve HBeAg seroconversion and even HBsAg disappearance than entecavir(ETV) drugs, which may be related to the functional activation of pDCs in the case of hepatitis and the function enhancement of pDCs during Peg-IFN-α therapy. This study was aimed at investigating the changes of pDCs frequency and function, and the expression of costimulatory molecules CD86 during Peg-IFN-αandentecavir(ETV) therapy.Meanwhile,investigators want to explore whether the decline of HBsAg and HBeAg resulted in recovery of CD86+pDC function, or recovery of CD86 + pDC function led to the decrease of HBsAg and HBeAg. Several studies demonstrated that HBsAg and HBeAg could damage pDC function, and the loss of HBsAg and HBeAg led to recovery of CD86+pDC function.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg and HBeAg positive for more than 6 months, HBVDNA detectable with ALT(alanine aminotransferase) level abnormal lasted for three months and at least time190 IU/L or liver puncture biopsy demonstrated apparent inflammation, never treated before enrolled.

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: the population in this study was composed of HBeAg positive chronic hepatitis B patients defined as HBsAg positive, HBeAg positive, and detectable HBVDNA load with ALT(alanine aminotransferase) level ≥190 U/L for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the change of pDC% | after treatment 24 weeks
  The host immune function will be evaluated by pDC. pDC% will be measured by flow cytometry after Pegylated Interferon α-2a and entecavir(ETV) Treatment 24 weeks.
the change of CD86+pDC% | after treatment 24 weeks
  CD86+pDC% will be measured by flow cytometry after Pegylated Interferon α-2a and entecavir(ETV) Treatment 24 weeks.
the change of mean fluorescence intensity of costimulatory molecules CD86(CD86-MFI) | after treatment 24 weeks
  mean fluorescence intensity of costimulatory molecules CD86(CD86-MFI) will be measured by flow cytometry after Pegylated Interferon α-2a and entecavir(ETV) Treatment 24 weeks.
the change of absolute molecular counting of costimulatory molecules CD86 | after treatment 24 weeks
  absolute molecular counting of costimulatory molecules CD86 (CD86-ABC) will be measured by flow cytometry after Pegylated Interferon α-2a and entecavir(ETV) Treatment 24 weeks.

SECONDARY OUTCOMES:
the change of HBVDNA levels (IU/ML) | after treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBV DNA levels
the change of ALT levels(U/L) | after treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by ALT levels
the change of AST levels(U/L) | after treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by AST levels
the change of HBsAg levels (IU/ML) | after treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBsAg levels
the change of HBeAg levels (IU/ML) | after treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBeAg levels

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China